CLINICAL TRIAL: NCT06696794
Title: Investigating the Efficacy and Safety of Neoadjuvant Intravesical Instillation of Mitomycin C Combined with En-bloc Surgery in Treating High-risk Non-muscle-invasive Bladder Cancer (NMIBC) Patients
Brief Title: Investigating the Efficacy and Safety of Neoadjuvant Intravesical Instillation of Mitomycin C in Treating High-risk NMIBC Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shaogang Wang (Other)
Responsible Party: Sponsor-Investigator, Shaogang Wang, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024TJCR012
Record Dates: First submitted 2024-11-17; First posted 2024-11-20 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-11

CONDITIONS: Non-Muscle-Invasive Bladder Cancer (NMIBC)
Keywords: high-risk non-muscle-invasive bladder cancer; neoadjuvant intravesical instillation; mitomycin C; en-bloc surgery
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — Mitomycin; Saline Solution

STUDY DESIGN:
Intervention Model Description: This was a double-blind, parallel-group, placebo-controlled, multicenter, prospective, randomized controlled Phase III clinical trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neoadjuvant intravesical instillation mitomycin C combined with en-bloc surgery (Experimental)
  Interventions: Drug: Mitomycin C (MMC)
- Neoadjuvant intravesical instillation normal saline combined with en-bloc surgery (Placebo Comparator)
  Interventions: Drug: Normal Saline (Placebo)

INTERVENTIONS:
Drug: Mitomycin C (MMC) — When administering neoadjuvant intravesical instillations, instruct the patient to lie flat on the treatment bed and cover with a waterproof pad. Disinfect the perineal area 2-3 times. Under sterile conditions, insert a catheter and drain the bladder of urine completely. Slowly instill the prepared instillation solution (mitomycin) into the bladder. If the patient experiences pain during the instillation, stop the infusion immediately, and continue when the pain subsides. If the patient still cannot tolerate it, discontinue the instillation treatment for this session. After the medication is instilled into the bladder, the catheter can be removed immediately or left in place. Instruct the patient to hold their urine for as long as possible under suitable conditions for 2 hours, and to change positions intermittently while the medication is retained in the bladder. The neoadjuvant intravesical instillation cycle is twice (one day and 4 h before en-bloc surgery）
  Arms: Neoadjuvant intravesical instillation mitomycin C combined with en-bloc surgery
Drug: Normal Saline (Placebo) — When administering neoadjuvant intravesical instillations, instruct the patient to lie flat on the treatment bed and cover with a waterproof pad. Disinfect the perineal area 2-3 times. Under sterile conditions, insert a catheter and drain the bladder of urine completely. Slowly instill the prepared instillation solution (Normal Saline) into the bladder. If the patient experiences pain during the instillation, stop the infusion immediately, and continue when the pain subsides. If the patient still cannot tolerate it, discontinue the instillation treatment for this session. After the medication is instilled into the bladder, the catheter can be removed immediately or left in place. Instruct the patient to hold their urine for as long as possible under suitable conditions for 2 hours, and to change positions intermittently while the medication is retained in the bladder. The neoadjuvant intravesical instillation cycle is twice (one day and 4 h before en-bloc surgery）
  Arms: Neoadjuvant intravesical instillation normal saline combined with en-bloc surgery

SUMMARY:
The goal of this clinical trial is to learn if neoadjuvant intravesical instillation of mitomycin C combined with en-bloc surgery works to treat high-risk non-muscle-invasive bladder cancer (NMIBC) patients. It will also learn about the safety of neoadjuvant intravesical instillation of mitomycin C. The main questions it aims to answer are:

Does neoadjuvant intravesical instillation of mitomycin C heighten the 1-year recurrence-free survival (RFS) rate for high-risk non-muscle-invasive bladder cancer (NMIBC) patients? What medical problems do participants have when taking neoadjuvant intravesical instillation of mitomycin C? Researchers will compare neoadjuvant intravesical instillation of mitomycin C to a placebo (normal saline) to see if neoadjuvant intravesical instillation of mitomycin C works to treat high-risk NMIBC.

Participants will:

Take neoadjuvant intravesical instillation of mitomycin C or a placebo twice，1 day and 4 hours before en-bloc surgery Visit the clinic once every 8 weeks for checkups and tests Keep track of the recurrence and progression of the tumor.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign an informed consent form, understand the study and are willing and able to follow and complete all trial procedures
2. Gender is not limited, age between 18 to 75 years old (inclusive of boundary values)
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
4. Previously confirmed non-muscle-invasive bladder cancer by imaging and pathology
5. In accordance with the "EAU Guidelines (2024 edition)" high-risk NMIBC patient danger grouping. All T1 HG/G3 and CIS patients except for the extremely high-risk group; Ta LG/G2 or T1G1, non-CIS with three risk factors; Ta HG/G3 or T1 LG, non-CIS with at least two risk factors; T1G2 non-CIS with at least one risk factor. (Risk factors: age > 70 years; multiple papillary tumors; tumor diameter > 3cm)
6. Participants are willing to provide the last cystoscopy biopsy specimen or specimens from the previous recurrence surgery (including paraffin blocks, paraffin-embedded sections, etc.)
7. The interval between previous anti-tumor treatments (chemotherapy, radiotherapy, immunotherapy) and the first administration of this trial is ≥6 weeks
8. Suitable organ function and hematopoietic function: Neutrophil count (NEUT ≥ 1.5 × 10^9/L; White blood cell count (WBC) ≥ 3.0 × 10^9/L; Platelet count ≥ 100 × 10^9/L; Hemoglobin ≥ 90g/L; Serum creatinine ≤ 1.5 times the upper limit of normal (ULN); AST and ALT ≤ 2.5 times ULN; Serum total bilirubin ≤ 1.5 times ULN; Activated partial thromboplastin time (APTT) ≤ 1.5 times ULN (except for patients on anticoagulant therapy)
9. Male participants must agree to use effective contraceptive measures during the treatment period and for at least 180 days after the last treatment, and must not donate sperm during this period; women of childbearing age must have a negative blood pregnancy test within 72 hours before the first new adjuvant instillation, and must agree to use effective contraceptive measures during the treatment period and for at least 180 days after en-bloc treatment

Exclusion Criteria:

1. The primary tumor is upper urinary tract urothelial carcinoma of the renal pelvis and ureter
2. Patients who have suffered from malignant tumors other than bladder urothelial carcinoma within 5 years before enrollment. However, the following patients are included (eligible for enrollment): ① Patients with locally low-risk prostate cancer (staging ≤T2b, Gleason score ≤7, and PSA ≤ 20ng/ml, with no recurrence after treatment as determined by follow-up PSA levels); ② Patients with low-risk prostate cancer (staging T1/T2a, Gleason score ≤7, and PSA ≤10ng/ml, in the observation phase without treatment; ③ Patients who meet other enrollment criteria but have very low risk of metastasis or death from malignant tumors, and who show no recurrence or metastasis after standard treatment, as confirmed by imaging and disease-specific tumor marker tests, such as fully treated carcinoma in situ of the cervix, basal or squamous cell skin cancer; in situ ductal carcinoma after treatment surgery, etc
3. Patients with active autoimmune diseases who have required systemic treatment (i.e., long-term use of corticosteroids or immunosuppressive drugs) within the past two years. Replacement therapy (such as thyroid hormone, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency) is excluded
4. Patients who are expected to have major surgery during the study period or who have undergone major surgery within 4 weeks before dosing and have not fully recovered
5. Any immune-related toxicity caused by previous cancer treatments has not recovered to ≤Grade 1 (except for Grade 2 endocrine disorders on stable dose steroid replacement therapy), and/or any other toxicity related to previous anti-cancer treatments (immune-related toxicity excluded) has not recovered to ≤Grade 2, except for alopecia
6. Patients who are seropositive for Human Immunodeficiency Virus (HIV) or have a history of HIV infection or other acquired immunodeficiency diseases
7. Patients who require long-term antiviral medication for hepatitis B or C, where hepatitis B (must meet both HBsAg positivity and HBV DNA ≥2000 IU/ml, excluding drug or other causes of hepatitis), hepatitis C (must meet both anti-HCV antibody positivity and HCV-RNA results greater than the lower limit of detection)
8. Uncontrolled stable systemic diseases, such as cardiovascular and cerebrovascular diseases, diabetes, etc
9. History of organ transplantation or stem cell transplantation
10. Heart failure (patients classified as NYHA Class III-IV according to the New York Heart Association)
11. Significant pulmonary disease (such as shortness of breath at rest or with mild activity or requiring oxygen for any reason)
12. Other underlying diseases judged by the investigator before the study that prevent the use of study medication or interfere with disease diagnosis, or have the potential to cause serious complications
13. Concurrent other serious infections before dosing
14. Alcohol dependence or a history of drug or substance abuse within the last year
15. A history of clear neurological or psychiatric disorders, such as epilepsy, dementia, poor compliance, or the presence of peripheral nervous system disorders
16. Pregnancy or breastfeeding, or expected to be pregnant or give birth during the trial period
17. Known allergy or intolerance to intravenous mitomycin and corresponding excipients
18. Patients whom the investigator deems unsuitable for the trial for other reasons

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
1-year recurrence-free survival rate | One year after randomization
  The one-year recurrence-free survival rate, as assessed by researchers, is defined as the proportion of patients who are free of tumor recurrence at one year after randomization. Recurrence is defined as any pathological level of urothelial carcinoma confirmed by cystoscopy and biopsy during the one-year follow-up period starting from the time of randomization.

SECONDARY OUTCOMES:
Progression free survival | Every eight weeks for one year and telephone follow-up every one year after one year until tumor progression and patient death from any cause, or five years after the end of the study.
  This was determined by cystoscopy and pathology every eight weeks for one year and telephone follow-up every one year after one year until tumor progression and patient death from any cause, or five years after the end of the study. Defined as the time between the start of randomization and progression of disease or death from any cause, whichever occurs first. Disease progression was defined as an increase in bladder tumors from Ta/T1 to T1/ T2 or larger, lymph node metastasis and distant metastasis, or an increase in tumor grade from low to high.
overall survival | up to 5 years after the end of the study.
  Telephone follow-up was conducted every 1 year after the start of randomization until death from any cause or 5 years after the end of the study.
Health-related quality of life | up to One year after discharge
  The health-related quality of life of the patients was assessed by EORTC QLQ-C30
Adverse event | up to Eight weeks after discharge
  Adverse events were coded using the International Dictionary of Medical Terms (MedDRA), and adverse events (TEAE) during treatment were aggregated by Systematic Organ Classification (SOC), Preferred term (PT), and NCI-CTCAE grading. The number, frequency and incidence of adverse events and drug-related adverse events of all subjects were counted. Make a list of adverse events. This is determined by interview, physical examination, as well as the patient's vital signs and laboratory tests.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The central Hospital of wuhan, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol